CLINICAL TRIAL: NCT00816166
Title: Phase III Study of Pharos Vitesse Neurovascular Stent System Compared to Best Medical Therapy for the Treatment of Ischemic Disease
Brief Title: VISSIT Intracranial Stent Study for Ischemic Therapy
Acronym: VISSIT
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Codman & Shurtleff (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VISSIT CA-2007-01; G080051
Record Dates: First submitted 2008-12-29; First posted 2008-12-31 (Estimated); Results first posted 2014-06-16 (Estimated); Last update posted 2015-02-20 (Estimated); Status verified 2015-02

CONDITIONS: Ischemic Stroke; Transient Ischemic Attack
Keywords: Ischemic stroke; Transient Ischemic Attack; Intracranial Stenting
MeSH Terms: conditions — Ischemic Stroke; Ischemic Attack, Transient | interventions — Aspirin; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stent Group (Experimental): Medical therapy + PHAROS Vitesse neurovascular stent ("Stent Group")
  Interventions: Device: Pharos Vitesse Neurovascular Stent System (Stent implantation) + Medical therapy (Aspirin and Clopidogrel)
- Medical Therapy Group (Active Comparator): Medical therapy alone ("Medical Therapy Group")
  Interventions: Drug: Aspirin and Clopidogrel (Medical therapy)

INTERVENTIONS:
Device: Pharos Vitesse Neurovascular Stent System (Stent implantation) + Medical therapy (Aspirin and Clopidogrel) — Implantation of one or more balloon-expandable Pharos Vitesse stents to treat neurovascular ischemic lesions + Medical therapy [Treatment with aspirin (81-325 mg daily for the duration of the study) and Clopidogrel (75 mg daily for first 3 months)]
  Other Names: Pharos Vitesse Neurovascular Stent System; Asprin; Clopidogrel; Plavix(r)
  Arms: Stent Group
Drug: Aspirin and Clopidogrel (Medical therapy) — Medical therapy alone [Treatment with aspirin (81-325 mg daily for the duration of the study) and Clopidogrel (75 mg daily for first 3 months)]
  Other Names: Aspirin; Clopidogrel; Plavix(r)
  Arms: Medical Therapy Group

SUMMARY:
The main objective of this study is to prospectively evaluate the safety, probable benefit, and effectiveness of the PHAROS Vitesse Neurovascular Stent System in a multicenter, randomized clinical trial.

A secondary objective of this study is to evaluate the impact of stenting in the neurovasculature to treat cerebral ischemia on other outcomes such as hospital length of stay, charges, and costs.

DETAILED DESCRIPTION:
1.1 Study Hypothesis Treatment of cerebral or retinal ischemia due to plaque in the neurovasculature using the PHAROS Vitesse Stent System plus medical therapy will provide additional clinical benefit over medical therapy alone.

1.2 Primary Effectiveness Endpoint

The primary effectiveness endpoint consists of a composite of the two following outcomes:

* Stroke in the same territory (distal to the target lesion) as the presenting event within 12 months of randomization
* Hard TIA in the same territory (distal to the target lesion) as the presenting event from day 2 through month 12 post-randomization

1.3 Safety Outcomes

Safety outcomes to be collected and reported as part of the overall risk-to-benefit profile for this device are:

* Stroke in any territory within 30 days of randomization
* Death from any cause within 30 days of randomization
* Hard TIA in any territory occurring after a 24 hour post-procedure stabilization period (days 2-30) since the recovery from anesthesia can mask accurate assessment of possible TIA symptoms.
* Intracranial hemorrhage within 30 days of randomization

1.4 Other Outcomes

* Stent Success - PHAROS Vitesse stent deployed across target lesion with residual stenosis 0-20%
* Percentage of Stent Group Subjects with any (symptomatic or asymptomatic) in-stent restenosis ≥ 70% confirmed by angiogram at 12 months
* Percentage of Stent Group Subjects with symptomatic in-stent restenosis ≥ 70% confirmed by angiogram at 12 months
* Percentage of Medical Therapy Group Subjects with interventional procedure (e.g., angioplasty or stent) at 12 months
* Comparison of NIHSS scores between treatment arms
* Comparison of mRS scores between treatment arms

ELIGIBILITY:
Inclusion Criteria:

1. Subject has at least one neurovascular lesion (70-99%) stenosis [internal carotid, middle cerebral, vertebral artery (C4-BA), and/or basilar artery] symptomatic with a hard TIA or stroke attributable to the territory of the lesion within the past 30 days. An intracranial tandem lesion (50-99%) stenosis may be treated if normal artery segment is sufficient length to avoid overlapping stents.
2. Target vessel diameter / lesion length measurements are within one of the below per angiogram:

   * Vessel diameter is ≥ 2.0 mm and < 2.5 mm / lesion length is ≤ 16 mm, or
   * Vessel diameter is ≥ 2.5 mm and < 3.0 mm / lesion length is ≤ 18 mm, or
   * Vessel diameter is ≥ 3.0 mm and < 4.5 mm / lesion length is ≤ 26 mm, or
   * Vessel diameter is ≥ 4.5 mm and ≤ 5.0 mm / lesion length is ≤ 31 mm
3. Subject has normal artery adjacent to each stenosis; diameter 2.0 mm - 5.0 mm
4. Subject age is 18-85 years
5. Life expectancy is at least 2 years
6. Subject 's mRS score is ≤ 3
7. Subject is available for study follow-up visits (e.g., lives within 3 hours of research center)
8. Subject is willing and cognitively able to provide Informed Consent (consent may be indicated verbally and signed by neutral witness if stroke has impaired hand or visual function)

Exclusion Criteria:

1. Subject has contraindications for balloon expandable stent, e.g.

   * Extreme tortuosity at, or proximal to, target lesion,
   * More than 2 lesions with > 50% stenosis (including vertebral ostia and common carotid disease),
   * Carotid or vertebral dissection
2. CT scan or MRI evidence of any of the following:

   * Intracranial hemorrhage of type PH1 or PH2
   * Subdural or epidural hemorrhage
   * Mass effect, or
   * Intracranial tumor (except small meningioma)
3. Subject has a previous stent in the territory of the target lesion(s)
4. Subject has a previous coil or clip placed in the territory of the target lesion within 6 months
5. Subject has a potential source of cardiac embolism requiring anticoagulation therapy (e.g., atrial fibrillation, intracardiac thrombus or vegetation, significant mitral stenosis, mechanical heart valve, congestive heart failure with EF <30%, or endocarditis)
6. Subject has concurrent intracranial pathology, e.g.

   * Moyamoya
   * Vasculitis documented by biopsy results
   * Ruptured Aneurysm
   * Unruptured aneurysm > 7mm
7. Subject has uncontrolled hypertension (systolic >185 mmHg or diastolic >110 mmHg)
8. Hemoglobin < 10 g/dL; platelet count < 100,000; or INR > 1.5 (e.g., use of warfarin)
9. Subject has an uncorrectable bleeding diathesis
10. Subject's neurological status is unstable and rapidly declining (NIHSS score increased > 4 points within 48 hours prior to randomization)
11. Subject has a contraindication for combination antithrombotic treatment (e.g., clopidogrel and aspirin) such as peptic ulcer disease
12. Subject history indicates high risk of non-compliance (e.g., substance abuse, psychosocial issues, etc.)
13. Subject has a known history contraindicating contrast dye or iodine (vs. sensitivity which can be safely controlled by antihistamine, steroid, etc.)
14. Subject is pregnant or plans to become pregnant in the next 12 months
15. Myocardial infarction within past 3 months
16. Treatment with tPA or other thrombolytic agent within 48 hours prior to randomization
17. Major surgery or trauma within 2 weeks prior to randomization
18. Enrollment in another investigational device or drug study that may confound the results

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2008-10; Primary Completion 2013-04 (Actual); Study Completion 2014-06 (Actual)

REFERENCES:
- [Background] Berkefeld J, Hamann GF, du Mesnil R, Kurre W, Steinmetz H, Zanella FE, Sitzer M. [Endovascular treatment for intracranial stenoses. A common statement by neurologists and neuroradiologists]. Nervenarzt. 2006 Dec;77(12):1444-55. doi: 10.1007/s00115-006-2182-z. German. PMID 17119891
- [Background] Chimowitz MI, Lynn MJ, Howlett-Smith H, Stern BJ, Hertzberg VS, Frankel MR, Levine SR, Chaturvedi S, Kasner SE, Benesch CG, Sila CA, Jovin TG, Romano JG; Warfarin-Aspirin Symptomatic Intracranial Disease Trial Investigators. Comparison of warfarin and aspirin for symptomatic intracranial arterial stenosis. N Engl J Med. 2005 Mar 31;352(13):1305-16. doi: 10.1056/NEJMoa043033. PMID 15800226
- [Background] Cruz-Flores S, Diamond AL. Angioplasty for intracranial artery stenosis. Cochrane Database Syst Rev. 2006 Jul 19;2006(3):CD004133. doi: 10.1002/14651858.CD004133.pub2. PMID 16856032
- [Background] Derdeyn CP, Chimowitz MI. Angioplasty and stenting for atherosclerotic intracranial stenosis: rationale for a randomized clinical trial. Neuroimaging Clin N Am. 2007 Aug;17(3):355-63, viii-ix. doi: 10.1016/j.nic.2007.05.001. PMID 17826637
- [Background] Fiorella D, Chow MM, Anderson M, Woo H, Rasmussen PA, Masaryk TJ. A 7-year experience with balloon-mounted coronary stents for the treatment of symptomatic vertebrobasilar intracranial atheromatous disease. Neurosurgery. 2007 Aug;61(2):236-42; discussion 242-3. doi: 10.1227/01.NEU.0000255521.42579.31. PMID 17762735
- [Background] Fiorella D, Woo HH. Emerging endovascular therapies for symptomatic intracranial atherosclerotic disease. Stroke. 2007 Aug;38(8):2391-6. doi: 10.1161/STROKEAHA.107.482752. Epub 2007 Jun 21. No abstract available. PMID 17585085
- [Derived] Zaidat OO, Fitzsimmons BF, Woodward BK, Wang Z, Killer-Oberpfalzer M, Wakhloo A, Gupta R, Kirshner H, Megerian JT, Lesko J, Pitzer P, Ramos J, Castonguay AC, Barnwell S, Smith WS, Gress DR; VISSIT Trial Investigators. Effect of a balloon-expandable intracranial stent vs medical therapy on risk of stroke in patients with symptomatic intracranial stenosis: the VISSIT randomized clinical trial. JAMA. 2015 Mar 24-31;313(12):1240-8. doi: 10.1001/jama.2015.1693. PMID 25803346

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened and enrolled at 27 sites worldwide (23 sites in the US and 4 sites outside of the US).
Pre-assignment Details: 125 consented,of which 112 were randomized.Of 112,110 were treated (64 Stent Arm & 46 Med Therapy [MT] Arm).Of 112, 111 met criteria & in analysis pop (58 Stent Arm & 53 MT Arm).During course of the study,of 59 randomized to Stent Arm,4 treated w/MT Only & 1 failed to meet eligibility & excluded, & of 53 randomized to MT Arm, 9 treated w/Stent+MT.
Groups:
- Stent Group: Medical therapy + PHAROS Vitesse neurovascular stent ("Stent Group")
  Pharos Vitesse Neurovascular Stent System (Stent implantation): Implantation of one or more balloon-expandable Pharos Vitesse stents to treat neurovascular ischemic lesions.
- Medical Therapy Group: Medical therapy alone ("Medical Therapy Group")
  Aspirin and Clopidogrel (Medical therapy): Treatment with aspirin (81-325 mg daily for the duration of the study) and Clopidogrel (75 mg daily for first 3 months)
Period: Overall Study
Arm/Group | Stent Group | Medical Therapy Group
Started | 59 (Of 59 randomized to Stent Arm, 4 were treated with Medical Therapy Only) | 53 (Of 53 randomized to Medical Therapy Arm, 9 were treated with Stent+Medical Therapy)
ITT Population (Met Eligibility) | 58 (Of 59 randomized to Stent Arm, 1 subject failed to meet eligibility and was excluded from the ITT) | 53
Completed | 49 | 41
Not Completed | 10 | 12
Not completed — Lost to Follow-up | 6 | 10
Not completed — Death | 4 | 2

BASELINE CHARACTERISTICS:
Population: Analyses were based on an Intent-to-Treat (ITT) population, defined ad enrolled subjects who met the inclusion/exclusion criteria and who were randomized post angiogram. Stent and medical Therapy Group subjects were analyzed to their ITT randomized group regardless of treatment received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Stent Group | Medical Therapy Group | Total
Number analyzed (Participants) | 58 | 53 | 111
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.8 (12.3) | 61.8 (12.8) | 61.8 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 21 | 38
  Male | 41 | 32 | 73
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 2 | 7
  Not Hispanic or Latino | 53 | 51 | 104
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 7 | 7 | 14
  Native Hawaiian or Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 5 | 9
  White | 42 | 38 | 80
  Unknown or Not Reported | 5 | 3 | 8
Region of Enrollment [Number; unit: participants]
  United States | 47 | 42 | 89
  China | 7 | 7 | 14
  Austria | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Successful Outcome: No Stroke or Hard TIA in the Same Territory Within 12 Months
Description: The primary effectiveness endpoint was a composite of the two following outcomes:
  * Stroke in the same territory (distal to the target lesion) as the presenting event within 12 months of randomization
  * Hard Transient Ischemic Attack (TIA) in the same territory (distal to the target lesion) as the presenting event from day 2 through month 12 post-randomization
  A subject was deemed to be a primary endpoint success if neither of these outcomes occurred.
  The Kaplan-Meier success rate at 12-months post-operatively was calculated with Kaplan-Meier time-to-event methodology, where the time variable for patients who were successful (no stroke within 12 months or hard TIA between 2 days and 12 months) was censored at the time of last follow-up, and the time variable for patients who were not successful (had a stroke within 12 months or hard TIA between 2 days and 12 months) was censored at the time of the first event (stroke with 12 months or hard TIA between 2 days and 12 months).
Time Frame: One Year
Population: Analyses were based on an intent-to-treat (ITT) population, defined as enrolled subjects who met the inclusion/exclusion criteria and who were randomized post angiogram. Stent and Medical Therapy Group subjects were analyzed according to their ITT randomized group regardless of treatment received.
Measure: Number (95% Confidence Interval); unit: percent probability
Arm/Group | Stent Group | Medical Therapy Group
Number analyzed (Participants) | 58 | 53
percent probability | 62.24 [48.15 to 73.15] | 83.68 [69.94 to 91.50]

ADVERSE EVENTS:
Time Frame: Adverse events were collect from time of baseline angiogram/stent procedure through subject end of study (either early termination or 12 month post procedure follow up visit)
Description: Adverse events collected and were summarized according to how they were reported by investigational sites
Arm/Group | Stent Group | Medical Therapy Group
Serious Adverse Events (participants affected / at risk) | 30/58 | 20/53
Other Adverse Events (participants affected / at risk) | 37/58 | 34/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stent Group (N=58) | Medical Therapy Group (N=53)
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Chest pain (Cardiac disorders) | 0 (0) | 2 (2)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Oedema peripheral (Cardiac disorders) | 0 (0) | 1 (1)
Syncope (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Endocrine disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Endocrine disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Completed suicide (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0)
Medical device pain (General disorders) | 0 (0) | 1 (1)
Neurological symptom (General disorders) | 1 (1) | 0 (0)
Stent malfunction (General disorders) | 1 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 2 (2)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Arterial restenosis (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 2 (2) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 2 (2) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 7 (7) | 4 (4)
Muscular weakness (Nervous system disorders) | 1 (1) | 0 (0)
Neurological symptom (Nervous system disorders) | 2 (2) | 0 (0)
Post procedural stroke (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 2 (2)
Vertebrobasilar insufficiency (Nervous system disorders) | 1 (1) | 0 (0)
Vision blurred (Nervous system disorders) | 1 (1) | 0 (0)
Visual field defect (Nervous system disorders) | 1 (1) | 0 (0)
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 3 (3) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Amputation (Surgical and medical procedures) | 1 (1) | 0 (0)
Carotid endarterectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Hip arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Artery dissection (Vascular disorders) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Intermittent claudication (Vascular disorders) | 1 (1) | 0 (0)
Migraine (Vascular disorders) | 0 (0) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Vascular disorders) | 2 (2) | 4 (5)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stent Group (N=58) | Medical Therapy Group (N=53)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 2 (2)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Haemoglobin decreased (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Chest discomfort (Cardiac disorders) | 0 (0) | 1 (1)
Chest pain (Cardiac disorders) | 0 (0) | 2 (2)
Coronary Artery Disease (Cardiac disorders) | 1 (1) | 1 (1)
Dizziness (Cardiac disorders) | 0 (0) | 1 (1)
Dizziness postural (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Oedema peripheral (Cardiac disorders) | 0 (0) | 1 (1)
Presyncope (Cardiac disorders) | 1 (1) | 0 (0)
Syncope (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 2 (2)
Diabetic neuropathy (Endocrine disorders) | 1 (1) | 0 (0)
Diabetic retinopathy (Endocrine disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Endocrine disorders) | 3 (3) | 0 (0)
Hypoglycaemia (Endocrine disorders) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 1 (1)
Retinal haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Visual field defect (Eye disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Barrett s oesophagus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 5 (5) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Dysphagia (Eye disorders) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Oropharyngeal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Post procedural diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 1 (1)
Lethargy (General disorders) | 0 (0) | 1 (1)
Localised oedema (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1)
Neurological complication associated with device (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Helicobacter infection (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Arterial restenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 6 (6) | 4 (4)
Phlebitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Procedural hypotension (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Procedural vomiting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood creatine increased (Investigations) | 1 (1) | 0 (0)
Blood glucose fluctuation (Investigations) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 1 (1) | 0 (0)
Blood potassium abnormal (Investigations) | 1 (1) | 0 (0)
Blood potassium decreased (Investigations) | 1 (1) | 0 (0)
Blood testosterone decreased (Investigations) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
Neurological examination abnormal (Investigations) | 0 (0) | 1 (1)
Radial pulse decreased (Investigations) | 0 (0) | 1 (1)
Red blood cell sedimentation rate increased (Investigations) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint dislocation (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Wrist fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 1 (1)
Cerebral artery stenosis (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Diabetic gastroparesis (Nervous system disorders) | 1 (1) | 0 (0)
Diplopia (Nervous system disorders) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 4 (5) | 3 (4)
Hemiparesis (Nervous system disorders) | 2 (2) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 2 (2) | 0 (0)
Neuralgia (Nervous system disorders) | 2 (3) | 0 (0)
Neurological symptom (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 3 (4) | 2 (2)
Post stroke depression (Nervous system disorders) | 2 (2) | 1 (1)
Procedural headache (Nervous system disorders) | 1 (1) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 1 (1)
VIIth nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Vision blurred (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Memory impairment (Psychiatric disorders) | 1 (1) | 1 (1)
Withdrawal syndrome (Psychiatric disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 1 (1) | 0 (0)
Post procedural haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal cyst (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 2 (2) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 5 (5) | 1 (2)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Breast Mass (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Radiation pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dry gangrene (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Cataract operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 1 (1) | 0 (0)
Artery dissection (Vascular disorders) | 2 (2) | 0 (0)
Contusion (Vascular disorders) | 1 (1) | 0 (0)
Epistaxis (Vascular disorders) | 1 (1) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 7 (9) | 7 (10)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)
Post procedural haematoma (Vascular disorders) | 3 (4) | 0 (0)
Post procedural haemorrhage (Vascular disorders) | 1 (1) | 1 (1)
Subclavian artery stenosis (Vascular disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Vascular disorders) | 2 (2) | 8 (12)
Vasospasm (Vascular disorders) | 4 (4) | 0 (0)
Venous thrombosis (Vascular disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Early termination of enrollment led to small numbers of subjects analyzed (less than 50% of the prospectively planned sample size). Various endpoints, subgroup and sensitivity analyses were not conducted because the study was not fully enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less